CLINICAL TRIAL: NCT03970512
Title: 30 Day Fitting of a New Toric Contact Lens
Brief Title: Apioc Toric/Spherical Single Vision Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lentechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEN004
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Refractive Errors
Keywords: contact lens; soft contact lens
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Apioc-A and Apioc-S Contact Lenses — Appropriately fit, document and dispense a new spherical and toric contact lens design worn for up to 35 days.

SUMMARY:
The Lentechs Apioc-S and Apioc-A contact lenses are made in an FDA-approved contact lens material indicated for single-vision and astigmatism. The novel lens design has a lenticular portion which is thicker than the optical portion of the lens. When applied to the eye, it is oriented in a superior position. Unlike contact lenses currently on the market, this innovative design improves lens stability by preventing lens rotation, and may improve tear flow behind the lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must provide written informed consent.
2. The subject must appear willing and able to adhere to the instructions set forth in this protocol.
3. At least 18 years of age and no more than 35 years of age.
4. ≤ 4.00 D of corneal astigmatism.
5. ≤ 4.00 D of refractive astigmatism.
6. Refractive error range +20.00 DS to -20.00 DS
7. Flat and steep keratometry readings within 40 to 50D.
8. Clear, healthy corneas with no irregular astigmatism.
9. Normal, healthy conjunctiva in both eyes.
10. Free of active ocular disease. Refractive error is permitted.
11. Be a current or former (within the last 12 months) contact lens wearer.
12. Best-corrected near and distance visual acuity better than or equal to 20/25.

Exclusion Criteria:

1. Irregular corneal astigmatism.
2. Presbyopia
3. Corneal scarring unless off line-of-site and well healed.
4. Pinguecula, pterygium, or other conjunctival thickness abnormalities that would interfere with soft contact lens wear.
5. Recent use of any ocular pharmaceutical treatments, including daily artificial tears, in the two weeks prior to the examination. Use of artificial tears less than 3 drops per week is permitted.
6. Systemic disease that would interfere with contact lens wear.
7. Currently pregnant or lactating (by self-report).
8. History of strabismus or eye movement disorder.
9. Active allergies that may inhibit contact lens wear.
10. Upper eyelid margin at or above the superior limbus.
11. History of ocular or lid surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 30 days
  LogMAR distance visual acuity

SECONDARY OUTCOMES:
Comfort | 30 days
  Contact Lens Dry Eye Questionnaire-8, scale range 0 minimum (better outcome) to 38 maximum (worse outcome).
Rotational Stability of Apioc-A | 30 days
  Clockwise or counter-clockwise rotation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Quinn, OD, MS, FAAO, Principal Investigator — Drs. Quinn, Foster & Associates; Jason R Miller, OD, MBA, Principal Investigator — Eyecare Professionals of Powell
Locations (2):
- United States (2):
  - Quinn Foster & Associates, Athens, Ohio
  - EyeCare Professionals of Powell, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No